CLINICAL TRIAL: NCT01976130
Title: Mechanisms of Lung Defense and Their Relationship With Airway Infection in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIBSP-MUC-2009-20
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Bacterial Infection in COPD
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bronchoscopy (Experimental): Procedure
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy

SUMMARY:
Study hypothesis:

Chronic Obstructive Pulmonary Disease (COPD) patients with chronic bacterial colonization have lower levels of mucins and antimicrobial peptides in their airways

DETAILED DESCRIPTION:
Main objective:

(1) To investigate the expression of mucins and antimicrobial peptides in patients with severe COPD and their relationship with the presence of bacteria in the airway

ELIGIBILITY:
Inclusion Criteria:

* COPD

Exclusion Criteria:

* Acute exacerbation in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Mucins in sputum | Day 1

SECONDARY OUTCOMES:
Antimicrobial peptides in sputum | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain